CLINICAL TRIAL: NCT02379247
Title: Phase I/II Study of BYL719 and Nab-Paclitaxel in Subjects With Locally Recurrent or Metastatic HER-2 Negative Breast Cancer
Brief Title: BYL719 and Nab-Paclitaxel in Locally Recurrent or Metastatic HER-2 Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Priyanka Sharma (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Priyanka Sharma, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719XUS06T
Record Dates: First submitted 2015-01-30; First posted 2015-03-04 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: HER-2 Negative; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose level 1 BYL-719/alpelisib (250mg)+Nab-paclitaxel (Experimental): BYL-719 (alpelisib): 250mg daily on day 1-28
  Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  Interventions: Drug: BYL-719 (alpelisib); Drug: Nab-paclitaxel
- Dose level 2 BYL-719 (alpelisib) (300mg)+Nab-paclitaxel (Experimental): BYL-719 (alpelisib): 300mg by mouth daily on day 1-28 of each 28 day cycle
  Nab-paclitaxel: 100mg/m2 given IV on days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  Interventions: Drug: BYL-719 (alpelisib); Drug: Nab-paclitaxel
- Dose level 3 BYL-719 (alpelisib) (350mg)+Nab-paclitaxel (Experimental): BYL-719 (alpelisib): 350mg by mouth daily on day 1-28 of each 28 day cycle
  Nab-paclitaxel: 100mg/m2 given IV on days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  Interventions: Drug: BYL-719 (alpelisib); Drug: Nab-paclitaxel
- BYL-719 (alpelisib) Dose Expansion (Experimental): BYL-719 (alpelisib): RP2D from Phase I by mouth daily on day 1-28 of each 28 day cycle
  Nab-paclitaxel: 100mg/m2 given IV on days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  Interventions: Drug: BYL-719 (alpelisib); Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: BYL-719 (alpelisib) — Oral PI3K inhibitor
  Other Names: Piqray
Drug: Nab-paclitaxel — IV taxane
  Other Names: Abraxane

SUMMARY:
Investigate the use of BYL719 (alpelisib) as combination therapy with Nab-Paclitaxel in locally recurrent or metastatic HER-2 negative breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer and the second leading cause of cancer related death in American women. Despite recent improvement in the treatment of breast cancer, 40,000 women still die each year in the US as a result of breast cancer. Chemotherapy (usually consisting of sequential single agent) remains the backbone of treatment for patients with HER-2 negative metastatic breast cancer. A majority of patients show an initial response to treatment, but all eventually show disease progression.

The purpose of this study is to determine the highest dose of BYL719 (alpelisib) combined with Nab-Paclitaxel that results in no serious side effects. The safety and effectiveness of BYL719 combined with Nab-Paclitaxel to treat patients with HER-2 negative metastatic breast cancer will be assessed, along with the determination of how long this drug combination will keep the disease from getting worse.

The study will be done in two parts:

Part 1 will determine the highest dose of BYL719 that is safe and tolerable to take in combination with Nab-Paclitaxel. Part 1 will be completed before Part 2 begins.

Part 2 will investigate whether taking BYL719 (at the dose determined in Part 1) + Nab-Paclitaxel is safe and effective for patients with HER-2 negative metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written Informed Consent Form.
2. Age ≥ 18 years
3. Histologically proven HER-2 negative breast cancer (HER-2 negative defined as HER IHC 0 or 1+ and/or HER-2 FISH negative); HER-2 negative breast cancer includes hormone positive (ER and/or PR positive) breast cancer and TNBC
4. HER-2 negative breast cancer that at the time of study entry is either stage III (locally advanced) disease not amenable to curative therapy or stage IV disease. Histological confirmation of recurrent/metastatic disease is encouraged but not required if clinical evidence of stage IV disease is available
5. Have measurable (defined as at least one lesion that can be accurately measured in at least one dimension [longest diameter to be recorded] with minimum lesion size of ≥ 2 cm on conventional measurement techniques or ≥ 1 cm on spiral computed tomography (CT) scan
6. No limitations to number of prior chemotherapies for metastatic disease. Treatment with prior taxanes (except Nab-Paclitaxel) is allowed as long as it has been 6 months or more since exposure to prior taxane.

   NOTE: For subjects who are, or who have previously received endocrine therapy for breast cancer, the treating investigator will decide how many days should pass between the last dose of endocrine therapy and the first dose of study treatment.
7. All patients should have received at least one line of chemotherapy in either the advanced or adjuvant setting and hormonal therapy (where appropriate)
8. Performance status of 2 or better as per ECOG criteria (See Appendix A for details)
9. Subject is able to swallow and retain oral medicines
10. Adequate marrow and organ function as defined below (labs must be performed within 14 days of subject registration)

    * Absolute neutrophil count ≥ 1500/uL
    * Platelets 100,000/uL (no transfusion allowed within 2 weeks)
    * Hemoglobin > 9 g/dL (which may be reached by transfusion)
    * Total bilirubin within normal range or ≤ 1.5X IULN if liver metastases are present or total bilirubin ≤ 3.0X IULN with direct bilirubin within normal range in subjects with well-documented Gilbert's Syndrome, which is defined as presence of unconjugated hyperbilirubinemia with normal results from CBC (including normal reticulocyte count and blood smear), normal liver function test results and absence of other contributing disease processes at the time of diagnosis
    * AST(SGOT)/ALT(SPGT) ≤ 2.5X IULN or ≤ 5X IULN if liver metastases are present
    * Serum creatinine ≤ 1.5X IULN
    * INR ≤ 1.5
    * Fasting plasma glucose ≤ 140 mg/dL or 7.8 mmol/L (NOTE: Fasting whole blood glucose testing is acceptable if fasting plasma glucose is not feasible.)
    * HBA1c ≤ 8%
    * Potassium, calcium (corrected for serum albumin) and magnesium within IULN
    * Serum Amylase < 2 x ULN and serum lipase within normal limits
11. IV bisphosphate and denosumab for bony metastatic disease will be allowed
12. Prior palliative radiation therapy to bony metastases is allowed. There should be a minimum of 14 days between the end of radiation treatment and start of study treatment
13. Subjects with previously treated brain metastases who are free of CNS symptoms and are > 3 months from treatment of brain metastases are eligible Subjects should be > 2 weeks from prior systemic chemotherapy for breast cancer AND should have recovered to Grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy prior to study entry NOTE: For subjects who are, or who have previously received endocrine therapy for breast cancer, the treating investigator will decide how many days should pass between the last dose of endocrine therapy and the first dose of study treatment.
14. Women of child bearing potential (WOCBP) and their partners must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. After confirmation of negative pregnancy test at screening, should a WOCBP become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician and the investigator immediately.

    * WOCBP are defined as any females (regardless of sexual orientation, having undergone tubal ligation, or remaining celibate by choice) who meet the following criteria:

      * Have not undergone a hysterectomy or bilateral oophorectomy OR
      * Have not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)

Exclusion criteria:

1. Subject has any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of drugs in this protocol or place the subject at undue risk for treatment complications
2. Subject is pregnant or lactating
3. Subject has previously been treated with Nab-Paclitaxel NOTE: Subjects who have had previous treatment with Nab-Paclitaxel will NOT be excluded if given in the adjuvant or neoadjuvant setting Only in the metastatic setting, will subjects previously treated with Nab-Paclitaxel be excluded from this trial. Exceptions may be made for subjects who discontinued treatment with a previous Nab-Paclitaxel inhibitor for reasons other than progression and as long as it has been > 12 months since discontinuation of the previous Nab-Paclitaxel. This exception will require prior approval from the study PI at KUMC.
4. Subject has inflammatory breast cancer
5. Subject has a known hypersensitivity to any of the excipients of Nab-Paclitaxel or BYL719/alpelisib
6. Subject has a concurrent malignancy or malignancy within 3 years of study enrollment (with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer)
7. Subject has clinically manifest diabetes mellitus or documented steroid-induced diabetes mellitus
8. Subject has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
9. Subject is classified into Child-Pugh class C
10. Subject has a known history of HIV infection (testing not mandatory)
11. Subject has active, uncontrolled infection
12. Subject has symptomatic/untreated CNS disease
13. Subject has ≥ Grade 2 peripheral neuropathy
14. Subject has active cardiac disease or a history of cardiac dysfunction including any of the following:

    * Unstable angina pectoris within 6 months prior to study entry
    * Symptomatic peritonitis
    * Documented myocardial infarction within 6 months prior to study entry
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    * Documented cardiomyopathy
    * Subject has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO)
    * Subject has any of the following cardiac conduction abnormalities
    * Ventricular arrhythmias except for benign premature ventricular contractions
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medicine
    * Conduction abnormality requiring a pacemaker
    * Other cardiac arrhythmia not controlled with medication
15. Subject has a QTcF > 480 msec on the screening ECG (using the QTcF formula)
16. Subject is currently receiving treatment with a medication that has a known risk to prolong the QT interval or induce Torsades de Pointes and the treatment cannot be discontinued or switched to a different medication prior to randomization
17. Subject has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects
18. Subject is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug or who have not fully recovered from side effects of such treatment
19. Subject is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A. The subject must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the start of treatment
20. Subject is currently receiving warfarin or other coumarin-derived anti-coagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
21. Subject has received previous treatment with a PI3K inhibitor. Exceptions may be made for subjects who discontinued treatment with a previous PI3K inhibitor for reasons other than toxicity or progression and as long as it has been > 12 months since discontinuation of the previous PI3K inhibitor. This exception will require prior approval from the study PI at KUMC.
22. Subjects who have received an investigational agent within 30 days OR within 5 half-lives of the investigational agent (whichever is shorter) prior to the possible enrollment date on this study.
23. Subject with history of acute within one year of study entry or past medical history of chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2022-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Sharma, MD, Principal Investigator — University of Kansas Medical Center
Locations (4):
- United States (4):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Sharma P, Abramson VG, O'Dea A, Nye L, Mayer I, Pathak HB, Hoffmann M, Stecklein SR, Elia M, Lewis S, Scott J, De Jong JA, Wang YY, Yoder R, Schwensen K, Finke K, Heldstab J, LaFaver S, Williamson SK, Phadnis MA, Reed GA, Kimler BF, Khan QJ, Godwin AK. Clinical and Biomarker Results from Phase I/II Study of PI3K Inhibitor Alpelisib plus Nab-paclitaxel in HER2-Negative Metastatic Breast Cancer. Clin Cancer Res. 2021 Jul 15;27(14):3896-3904. doi: 10.1158/1078-0432.CCR-20-4879. Epub 2021 Feb 18. PMID 33602685

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 BYL-719/Alpelisib (250mg)+Nab-paclitaxel: BYL-719 (alpelisib): 250mg daily on day 1-28
  Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  BYL-719 (alpelisib): Oral PI3K inhibitor
  Nab-paclitaxel: IV taxane
- Dose Level 2 BYL-719 (Alpelisib) (300mg)+Nab-paclitaxel: BYL-719 (alpelisib): 300mg by mouth daily on day 1-28 of each 28 day cycle
  Nab-paclitaxel: 100mg/m2 given IV on days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  BYL-719 (alpelisib): Oral PI3K inhibitor
  Nab-paclitaxel: IV taxane
- Dose Level 3 BYL-719 (Alpelisib) (350mg)+Nab-paclitaxel: BYL-719 (alpelisib): 350mg by mouth daily on day 1-28 of each 28 day cycle
  Nab-paclitaxel: 100mg/m2 given IV on days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  BYL-719 (alpelisib): Oral PI3K inhibitor
  Nab-paclitaxel: IV taxane
- BYL-719 (Alpelisib) Dose Expansion: BYL-719 (alpelisib): RP2D from Phase I by mouth daily on day 1-28 of each 28 day cycle
  Nab-paclitaxel: 100mg/m2 given IV on days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day)
  BYL-719 (alpelisib): Oral PI3K inhibitor
  Nab-paclitaxel: IV taxane
Period: Overall Study
Arm/Group | Dose Level 1 BYL-719/Alpelisib (250mg)+Nab-paclitaxel | Dose Level 2 BYL-719 (Alpelisib) (300mg)+Nab-paclitaxel | Dose Level 3 BYL-719 (Alpelisib) (350mg)+Nab-paclitaxel | BYL-719 (Alpelisib) Dose Expansion
Started | 3 | 3 | 7 | 30
Completed | 3 | 3 | 7 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 2 BYL-719/Alpelisib (300mg)+Nab-paclitaxel: BYL-719 (alpelisib): 300mg daily on day 1-28 Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day) BYL-719 (alpelisib): Oral PI3K inhibitor Nab-paclitaxel: IV taxane
- Dose Level 3 BYL-719/Alpelisib (350mg)+Nab-paclitaxel: BYL-719 (alpelisib): 350mg daily on day 1-28 Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day) BYL-719 (alpelisib): Oral PI3K inhibitor Nab-paclitaxel: IV taxane
- BYL-719/Alpelisib Dose Expansion: BYL-719 (alpelisib): RP2D from Phase I by mouth daily on day 1-28 of each 28 day cycle Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day) BYL-719 (alpelisib): Oral PI3K inhibitor Nab-paclitaxel: IV taxane
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 BYL-719/Alpelisib (250mg)+Nab-paclitaxel | Dose Level 2 BYL-719/Alpelisib (300mg)+Nab-paclitaxel | Dose Level 3 BYL-719/Alpelisib (350mg)+Nab-paclitaxel | BYL-719/Alpelisib Dose Expansion | Total
Number analyzed (Participants) | 3 | 3 | 7 | 30 | 43
Age, Continuous [Median (Full Range); unit: years] | 61 [41 to 65] | 61 [51 to 62] | 59 [52 to 68] | 54 [34 to 72] | 55 [34 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 30 | 43
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 7 | 30 | 43
Metastatic disease subtype [Count of Participants; unit: Participants] — Estrogen receptor and progesterone receptor positivity was defined as ≥10% by immunohistochemistry. HER2 positivity was defined per 2013 ASCO/CAP guidelines (Wolff et al, J Clin Oncol 2013;31(31):3997-4013. Triple negativity was defined as estrogen receptor negative, progesterone receptor negative, and HER2 negative.
  Participants
    Estrogen receptor and/or progesterone receptor positive | 1 | 2 | 4 | 23 | 30
    Triple-negative | 2 | 1 | 3 | 7 | 13
Measurable disease [Count of Participants; unit: Participants] — Presence of measurable disease according to RECIST version 1.1
  Participants | 3 | 3 | 7 | 30 | 43
Visceral disease [Count of Participants; unit: Participants] — Presence of at least one visceral metastatic site
  Participants
    Present | 3 | 3 | 6 | 24 | 36
    Absent | 0 | 0 | 1 | 6 | 7
Prior lines of chemotherapy for metastatic disease [Count of Participants; unit: Participants] — Number of prior lines of chemotherapy for metastatic disease.
  Participants
    0 | 0 | 1 | 2 | 7 | 10
    1 | 3 | 2 | 3 | 12 | 20
    ≥2 | 0 | 0 | 2 | 11 | 13
Prior taxane [Count of Participants; unit: Participants] — Prior receipt of a taxane, and in what treatment setting(s) a taxane was received.
  Participants
    Neoadjuvant or adjuvant | 2 | 2 | 5 | 17 | 26
    Metastatic only | 1 | 0 | 0 | 6 | 7
    Neoadjuvant or adjuvant AND metastatic | 0 | 0 | 0 | 3 | 3
    None | 0 | 1 | 2 | 4 | 7
Prior CDK4/6 inhibitor [Count of Participants; unit: Participants] — Prior receipt of any CDK4/6 inhibitor
  Participants
    Yes | 1 | 0 | 0 | 11 | 12
    No | 2 | 3 | 7 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose (RP2D) of BYL-719 (Alpelisib) + Nab-paclitaxel to be Used in Combination to Treat Advanced HER2-negative Breast Cancer
Description: Phase I was a 3+3 dose escalation design (three dose levels of alpelisib: 250mg, 300mg, and 350mg orally once daily, continuous dosing) with dose-limiting toxicities (DLT) assessed during the first treatment cycle. If two or more of the six patients experienced a dose-limiting toxicity, dosing escalation would cease and maximum tolerated dose (MTD) would be reached. RP2D was the next lower dose at which <1/6 subjects experienced a DLT.
Time Frame: 12 months
Measure: Number; unit: mg
Groups:
- Phase I: All patients in phase I, across all three dose levels of BYL-719 (alpelisib) + nab-paclitaxel
Arm/Group | Phase I
Number analyzed (Participants) | 13
mg | 350

2. Primary Outcome: Phase II: Overall Response Rate (ORR) of Subjects Treated at the Recommended Phase II Dose (RP2D)
Description: ORR includes complete response (CR) plus partial response (PR). As evaluated per RECIST version 1.1.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Participants Treated at the RP2D: Participants who were treated at the RP2D (350 mg BYL-719/alpelisib + 100 mg/m2 nab-paclitaxel) in either phase I or phase II.
Arm/Group | Participants Treated at the RP2D
Number analyzed (Participants) | 33
Participants | 17

3. Secondary Outcome: Clinical Benefit Rate (CBR) at 16 Weeks of Study Treatment
Description: CBR includes complete response (CR), partial response (PR), plus stable disease (SD) ≥16 weeks. As evaluated per RECIST version 1.1.
Time Frame: 16 weeks
Population: Per protocol the endpoint of CBR at 16 weeks is to be reported for all participants in phase I and phase II who were evaluable for response, thus participants from all assigned dose levels are combined for this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- All Evaluable Participants: All participants in phase I and phase II who were evaluable for response (i.e. received at least one cycle of study treatment)
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 42
Participants | 35

4. Secondary Outcome: Pharmacokinetics of BYL-719 (Alpelisib) When Administered With Nab-paclitaxel
Description: Area under the curve (AUC): sampling pre-dose and 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-alpelisib dose
Time Frame: In cycle 1 day 1, from prior to alpelisib dosing through 8 hours after alpelisib dosing
Population: Pharmacokinetic measures were assessed only among participants in phase I.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Dose Level 1: Participants assigned to dose level 1 BYL-719/Alpelisib (250mg)+Nab-paclitaxel
- Dose Level 2: Participants assigned to Dose Level 2 BYL-719/Alpelisib (300mg)+Nab-paclitaxel
- Dose Level 3: Participants in phase I assigned to dose level 3 BYL-719/Alpelisib (350mg)+Nab-paclitaxel
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 3 | 3 | 7
h*ng/mL | 6846 (3410) | 12436 (6174) | 13359 (5798)

5. Secondary Outcome: Pharmacokinetics of (Total) Nab-paclitaxel When Administered With BYL-719 (Alpelisib)
Description: Area under the curve (AUC): sampling pre-dose and 1.5, 2, 2.5, 3, 3.5, 4, and 6 hours post-alpelisib dose
Time Frame: In cycle 1 day 1, from prior to alpelisib dosing through 8 hours after alpelisib dosing
Population: Pharmacokinetic measures were assessed only among participants in phase I. One phase I participant assigned to the 350 mg BYL-719 (alpelisib) dose level did not have an end-of-infusion sample for paclitaxel measurement. Data are based on 12 participants.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 3 | 3 | 6
h*ng/mL | 8488 (1537) | 9938 (1735) | 6979 (2492)

6. Secondary Outcome: Progression-free Survival (PFS) and Overall Survival (OS)
Description: PFS was defined as the time in months from the date of enrollment to the date of progression or death, whichever was earlier. OS was defined as the time in months from the date of enrollment to death as a result of any cause. Survival curves were assessed by the Kaplan-Meier method.
Time Frame: 36 months
Population: Per protocol the endpoints of PFS and OS are to be reported for all participants in phase I and phase II who were evaluable for response, thus participants from all assigned dose levels are combined for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 42
months
  Progression-free survival | 8.7 [5.5 to 11.9]
  Overall survival | 18.5 [9.6 to 27.4]

7. Other Pre Specified Outcome: Correlation of PIK3CA Mutation With Clinical Benefit Rate
Description: Comparison of clinical benefit rate between participants with and without PIK3CA mutation in tumor tissue and/or circulating tumor DNA. Clinical benefit rate includes complete response (CR), partial response (PR), plus stable disease (SD) ≥16 weeks, as evaluated per RECIST version 1.1. Tumor DNA was isolated from archived formalin-fixed, paraffin-embedded tumor tissue (primary or metastatic site) and subjected to next-generation sequencing for assessment of PIK3CA mutation using ONCOReveal Multi-Cancer Panel (Pillar Biosciences). Circulating tumor DNA was isolated from pre-treatment plasma samples and subjected to next-generation sequencing for assessment of PIK3CA mutation using FoundationOne CDx testing or ONCOReveal Multi-Cancer Panel.
Time Frame: 24 months
Population: Among 42 participants evaluable for response, 17 had PIK3CA mutation in tumor tissue and/or circulating tumor DNA, while 25 did not. Clinical benefit rate was assessed among participants with PIK3CA mutation separately from participants without PIK3CA mutation for the purpose of correlating clinical benefit rate with PIK3CA mutation status. Per protocol the analysis is reported for all participants evaluable for response, thus participants from all dose levels are combined for this analysis.
Measure: Number; unit: participants
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 42
participants
  PIK3CA mutation present: number analyzed (Participants) | 17
  PIK3CA mutation present | 17
  PIK3CA mutation absent: number analyzed (Participants) | 25
  PIK3CA mutation absent | 17

ADVERSE EVENTS:
Time Frame: For each participant, treatment-related adverse events were collected from start of study treatment until 30 days after the participant's last dose of study treatment, assessed up to 174 weeks, whichever came first. All-cause mortality was collected from start of study treatment through October 16, 2019 (data cutoff date).
Description: Adverse events (serious and non-serious) of all grades, definitely related/probably related/possibly related to study treatment, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Patients were systematically evaluated for toxicity at each visit.
Groups:
- Dose Level 1 BYL-719/Alpelisib (250mg)+Nab-paclitaxel: BYL-719 (alpelisib): 250mg daily on day 1-28 of each 28 day cycle Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day) BYL-719 (alpelisib): Oral PI3K inhibitor Nab-paclitaxel: IV taxane
- Dose Level 2 BYL-719/Alpelisib (300mg)+Nab-paclitaxel: BYL-719 (alpelisib): 300mg daily on day 1-28 of each 28 day cycle Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day) BYL-719 (alpelisib): Oral PI3K inhibitor Nab-paclitaxel: IV taxane
- Dose Level 3 BYL-719/Alpelisib (350mg)+Nab-paclitaxel: BYL-719 (alpelisib): 350mg daily on day 1-28 of each 28 day cycle Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day) BYL-719 (alpelisib): Oral PI3K inhibitor Nab-paclitaxel: IV taxane
- BYL-719 (Alpelisib) Dose Expansion: BYL-719 (alpelisib): RP2D from Phase I by mouth daily on day 1-28 of each 28 day cycle Nab-paclitaxel: 100mg/m2 IV days 1, 8, 15 of each 28 day cycle (Window for Nab-paclitaxel is +/- 1 day) BYL-719 (alpelisib): Oral PI3K inhibitor Nab-paclitaxel: IV taxane
Arm/Group | Dose Level 1 BYL-719/Alpelisib (250mg)+Nab-paclitaxel | Dose Level 2 BYL-719/Alpelisib (300mg)+Nab-paclitaxel | Dose Level 3 BYL-719/Alpelisib (350mg)+Nab-paclitaxel | BYL-719 (Alpelisib) Dose Expansion
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 5/7 | 19/30
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/7 | 0/30
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 28/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 BYL-719/Alpelisib (250mg)+Nab-paclitaxel (N=3) | Dose Level 2 BYL-719/Alpelisib (300mg)+Nab-paclitaxel (N=3) | Dose Level 3 BYL-719/Alpelisib (350mg)+Nab-paclitaxel (N=7) | BYL-719 (Alpelisib) Dose Expansion (N=30)
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 6 | 19
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3 | 7 | 19
Nausea (Gastrointestinal disorders) | 3 | 2 | 3 | 20
Fatigue (General disorders) | 1 | 3 | 5 | 18
Peripheral neuropathy (Nervous system disorders) | 2 | 3 | 3 | 17
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 16
Electrolyte imbalance (Investigations) | 2 | 3 | 5 | 12
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 15
Mucositis (Gastrointestinal disorders) | 1 | 2 | 4 | 14
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 3 | 14
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 16
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 14
Infection (Infections and infestations) | 0 | 3 | 2 | 8
Edema (General disorders) | 0 | 2 | 3 | 7
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 8
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 7
Liver enzyme increase (Hepatobiliary disorders) | 1 | 1 | 1 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 6
Dry skin/mouth (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 5
Weight loss (Metabolism and nutrition disorders) | 0 | 1 | 2 | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 6 — Grade 3 generalized muscle weakness (n=1); grade 2 muscle weakness lower limb (n=2); grade 1 events (n=1 each): muscle weakness lower limb, left arm pain, generalized muscle weakness, and toe pain.
Creatinine imbalance (Renal and urinary disorders) | 0 | 1 | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Watering eyes (Eye disorders) | 0 | 1 | 0 | 3
Blurred vision (Eye disorders) | 0 | 0 | 0 | 3
Decreased lymphocyte count (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3
Dry eyes (Eye disorders) | 0 | 0 | 0 | 3
Fever (Infections and infestations) | 0 | 0 | 0 | 3
Gait disturbance (Nervous system disorders) | 0 | 1 | 1 | 1
Gastrointestinal - other (Gastrointestinal disorders) | 0 | 0 | 2 | 1 — Grade 2 colitis (n=1); grade 1 stomach tightness (n=1); and grade 1 unspecified gastrointestinal disorder (n=1).
Headache (Nervous system disorders) | 0 | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT02379247/Prot_SAP_000.pdf